CLINICAL TRIAL: NCT06766123
Title: Outcomes of Coronary Artery Bypass Grafting in Israeli Jews and Arabs
Status: Completed | Type: Observational
Sponsor: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Dror B. Leviner, Director of advanced cardiac surgery Department of cardiac surgery Carmel medical center, Technion, Israel Institute of Technology
Other Study IDs: CMC 21-175
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: CABG; Ethnic Group

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arab ethnicity: All Arab patients undergoing isolated CABG
  Interventions: Procedure: CABG
- Jew ethnicity: All Jew patients undergoing isolated CABG
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — All patients underwent isolated CABG and retrospectively followed to asses ethnic disparities

SUMMARY:
Retrospective study of adult patients with multivessel disease undergoing isolated CABG in three centers between January 1st, 2009, and December 31st, 2023. The primary outcome was a composite of major adverse cardiac and cerebrovascular events (MACCE). Patients were grouped according to their ethnic origin, Arabs and Jews.

ELIGIBILITY:
Inclusion Criteria:

* isolated CABG

Exclusion Criteria:

* members of different HMO

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing isolated CABG at Carmel medical center, Beilinson medical center and Soroka medical center at Israel
Sampling Method: Non-Probability Sample
Enrollment: 7067 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
MACCE | through study completion, a median of 78 months

SECONDARY OUTCOMES:
Mortality | through study completion, a median of 78 months
MI | through study completion, a median of 78 months
CVA | through study completion, a median of 78 months
repeat revascularization | through study completion, a median of 78 months
utilization of multi-arterial grafting | through study completion, a median of 78 months